CLINICAL TRIAL: NCT01627288
Title: Integrated Dose Escalation for Advanced, Localized Gynecologic Cancer (The IDEAL - GYN Trial)
Acronym: IDEAL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00033820
Record Dates: First submitted 2012-06-21; First posted 2012-06-25 (Estimated); Results first posted 2020-03-10 (Actual); Last update posted 2021-02-08 (Actual); Status verified 2021-02

CONDITIONS: Cancer of the Cervix; Cervical Neoplasms
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Boost Radiation: Dose Level 1 (Experimental): 2.4 Gy X 25 fractions = 60 Gy
  Interventions: Radiation: Boost radiation
- Boost Radiation: Dose level 2 (Experimental): 2.6 Gy X 25 fractions = 65 Gy
  Interventions: Radiation: Boost radiation
- Boost Radiation: Dose level 3 (Experimental): 2.8 Gy x 25 fractions = 70 Gy
  Interventions: Radiation: Boost radiation
- Experimental: Boost Radiation Dose Level 0 (Experimental): If the 2 dose limiting toxicities are documented at dose level 1, therapy will be de-escalated to Dose level 0 defined below.
  Dose level 0: 2.2 Gy X 25 fractions = 55 Gy
  Interventions: Radiation: Boost radiation

INTERVENTIONS:
Radiation: Boost radiation — Many studies have utilized a sequential boost to deliver a total dose of 55 - 60 Gy to the pelvic sidewall (covering the lower pelvic lymph nodes), including 8-10 Gy that is usually delivered with brachytherapy (1-3). This study treatment plan will escalate the dose to pelvic and para-aortic nodal disease from 60 Gy in 2.4 Gy per fraction to 70Gy in 2.8 Gy per fraction in 3 dose cohorts, using an integrated boost technique utilizing the same number of fractions for all cohorts (25 fractions) while the elective volumes are held constant at 45Gy

SUMMARY:
The purpose of this study is to determine the maximum tolerated dose of integrated boost radiation therapy when given with concurrent chemotherapy (cisplatin).

ELIGIBILITY:
Inclusion Criteria:

* Biopsy confirmed malignancy of the gynecologic tract
* Involved pelvic or para-aortic lymph nodes
* Treatment plan to include delivery of concurrent chemoradiotherapy.
* Good performance status
* Negative pregnancy test in women of child-bearing potential
* Signed study-specific informed consent
* Lab results within study specific limits

Exclusion Criteria:

* Prior radiation to the abdomen or pelvis
* A history of Scleroderma or Inflammatory bowel disease
* Contraindication to chemotherapy or radiation

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2012-06-04 (Actual); Primary Completion 2018-11-16 (Actual); Study Completion 2019-11-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Junzo Chino, MD, Principal Investigator — Duke Cancer Center/Radiation Oncology
Locations (1):
- Radiation Oncology, DUMC, Durham, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Boost Radiation Dose Level 0: If the 2 dose limiting toxicities are documented at dose level 1, therapy will be de-escalated to Dose level 0 defined below.
  Dose level 0: 2.2 Gy X 25 fractions = 55 Gy
Period: Overall Study
Arm/Group | Boost Radiation: Dose Level 1 | Boost Radiation: Dose Level 2 | Boost Radiation: Dose Level 3 | Boost Radiation Dose Level 0
Started | 3 | 3 | 6 | 0
Completed | 3 | 3 | 6 | 0
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: No subjects were reduced to Boost Radiation Level 0
Groups:
- Total: Total of all reporting groups
Arm/Group | Boost Radiation: Dose Level 1 | Boost Radiation: Dose Level 2 | Boost Radiation: Dose Level 3 | Boost Radiation Dose Level 0 | Total
Number analyzed (Participants) | 3 | 3 | 6 | 0 | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 3 | 2 | 6 | 0 | 11
  >=65 years | 0 | 1 | 0 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 6 | 0 | 12
  Male | 0 | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 3 | 3 | 6 | 0 | 12
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 2 | 1 | 0 | 0 | 3
  White | 1 | 2 | 6 | 0 | 9
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 3 | 3 | 6 |  | 12

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose of Integrated Boost Radiation Therapy, Administered With IMRT Technique With Concurrent Chemotherapy (Cisplatin).
Description: Concurrent radiation therapy and chemotherapy is the standard of care for node positive cervical cancer. While there are several acceptable means to boost the disease in the low pelvis (i.e. brachytherapy, IMRT, or external beam), there is limited research into boosting gross disease in the pelvis or para-aortic region. This protocol is designed to determine the maximum tolerated dose of treating tumor bearing regions within the abdomen and pelvis, using an integrated boost technique and concurrent chemotherapy.
Time Frame: During RT to 6 weeks post RT
Measure: Number; unit: Gray (Gy)
Groups:
- Treatment Arm: Participants received increasing doses of Radiation at 12.4 Gy X 25 fractions = 60 Gy (N=3), 2.6 Gy X 25 fractions = 65 Gy (N=6), or 2.8 Gy x 25 fractions = 70 Gy (N=12).
Arm/Group | Treatment Arm
Number analyzed (Participants) | 12
Gray (Gy) | 70

2. Secondary Outcome: Time to Local-regional Control With Integrated Boost Radiation Therapy (TTLR)
Description: Local-regional control is defined as local control without any nodal recurrence.
Time Frame: 3 years following treatment
Measure: Mean (Standard Deviation); unit: years
Groups:
- Combined Treatment Arms: Participants received increasing doses of Radiation at 12.4 Gy X 25 fractions = 60 Gy (N=3), 2.6 Gy X 25 fractions = 65 Gy (N=3), or 2.8 Gy x 25 fractions = 70 Gy (N=6).
- Boost Radiation: Dose Level 1 (60 Gy): Dose level 1 consists of a total 60Gy given in 2.4 Gy per fraction
- Boost Radiation: Dose Level 2 (65): Dose level 2 consists of a total 65Gy given in 2.6 Gy per fraction
- Boost Radiation: Dose Level 3 (70Gy): Dose level 3 consists of a total 70Gy given in 2.8 Gy per fraction
Arm/Group | Combined Treatment Arms | Boost Radiation: Dose Level 1 (60 Gy) | Boost Radiation: Dose Level 2 (65) | Boost Radiation: Dose Level 3 (70Gy)
Number analyzed (Participants) | 12 | 3 | 3 | 6
years | 1.5 (0.1) | NA (NA) — the value could not be calculated due to no events | 0.65 (NA) — the value could not be calculated due to too few events | 1.52 (0.04)

3. Secondary Outcome: Time to Distant Recurrence (TTDR)
Time Frame: 3 years after treatment
Measure: Mean (Standard Deviation); unit: years
Groups:
- Boost Radiation: Dose Level 2 (65): Dose level 1 consists of a total 65Gy given in 2.6 Gy per fraction
- Boost Radiation: Dose Level 3 (70Gy): Dose level 1 consists of a total 70Gy given in 2.8 Gy per fraction
Arm/Group | Combined Treatment Arms | Boost Radiation: Dose Level 1 (60 Gy) | Boost Radiation: Dose Level 2 (65) | Boost Radiation: Dose Level 3 (70Gy)
Number analyzed (Participants) | 12 | 3 | 3 | 6
years | 1.4 (0.1) | NA (NA) — the value could not be calculated due to no events | 1.2 (NA) — the value could not be calculated due to too few events | 1.29 (0.22)

4. Secondary Outcome: Disease Free Survival (DFS)
Time Frame: 3 years after treatment
Measure: Mean (Standard Deviation); unit: years
Arm/Group | Combined Treatment Arms | Boost Radiation: Dose Level 1 (60 Gy) | Boost Radiation: Dose Level 2 (65) | Boost Radiation: Dose Level 3 (70Gy)
Number analyzed (Participants) | 12 | 3 | 3 | 6
years | 1.3 (0.1) | 0.85 (NA) — the value could not be calculated due to too few events | 1.05 (0.23) | 1.34 (0.2)

5. Secondary Outcome: Overall Survival (OS)
Time Frame: 3 years after treatment
Measure: Mean (Standard Deviation); unit: years
Arm/Group | Combined Treatment Arms | Boost Radiation: Dose Level 1 (60 Gy) | Boost Radiation: Dose Level 2 (65) | Boost Radiation: Dose Level 3 (70Gy)
Number analyzed (Participants) | 12 | 3 | 3 | 6
years | 1.6 (0.1) | 0.85 (NA) — the value could not be calculated due to too few events | 1.08 (NA) — the value could not be calculated due to too few events | 1.7 (NA) — the value could not be calculated due to too few events

6. Secondary Outcome: Number of Participants With Acute Dose Limiting Toxicities (DLT)
Description: Acute DLT will be defined based on the side effects inherent from radiation therapy for gynecologic cancers, including effects on bowel, bladder, and skin.Since integrated radiation dose escalation is unlikely to substantially affect the hematopoietic system, only non-hematologic, grade 3-4, acute toxicity will be considered the primary dose-limiting toxicity (acute DLT). Dose limiting toxicity will include any of the following during treatment or within 6 weeks of completion: Acute Grade 3-4 enteritis or proctitis, Acute Grade 3-4 bladder toxicity, Acute Grade 4 dermatologic toxicity.
Time Frame: 6 weeks following treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Combined Treatment Arms | Boost Radiation: Dose Level 1 (60 Gy) | Boost Radiation: Dose Level 2 (65) | Boost Radiation: Dose Level 3 (70Gy)
Number analyzed (Participants) | 12 | 3 | 3 | 6
Participants | 1 | 0 | 0 | 1

7. Secondary Outcome: Number of Participants With Late Dose Limiting Toxicities (DLT)
Description: Late DLTs will be defined at grade 3-4 GI or GU toxicity with onset after 6 weeks of treatment.
Time Frame: 3 years following treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Combined Treatment Arms | Boost Radiation: Dose Level 1 (60 Gy) | Boost Radiation: Dose Level 2 (65) | Boost Radiation: Dose Level 3 (70Gy)
Number analyzed (Participants) | 12 | 3 | 3 | 6
Participants | 1 | 0 | 0 | 1

ADVERSE EVENTS:
Time Frame: 3 years
Groups:
- Dose Level 1: Participants received increasing doses of Radiation at 12.4 Gy X 25 fractions = 60 Gy (N=3)
- Dose Level 2: 2.6 Gy X 25 fractions = 65 Gy (N=3),
- Dose Level 3: 2.8 Gy x 25 fractions = 70 Gy (N=6)
Arm/Group | Dose Level 1 | Dose Level 2 | Dose Level 3
All-Cause Mortality (participants affected / at risk) | 1/3 | 1/3 | 1/6
Serious Adverse Events (participants affected / at risk) | 2/3 | 0/3 | 1/6
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 6/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dose Level 1 (N=3) | Dose Level 2 (N=3) | Dose Level 3 (N=6)
Nausea (Gastrointestinal disorders) | 1 | 0 | 0
Rectal necrosis (Gastrointestinal disorders) | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypokalemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Urinary fistula (Renal and urinary disorders) | 0 | 0 | 1
Urinary tract obstruction (Renal and urinary disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dose Level 1 (N=3) | Dose Level 2 (N=3) | Dose Level 3 (N=6)
Anemia (Blood and lymphatic system disorders) | 1 | 1 | 3
Colitis (Gastrointestinal disorders) | 1 | 0 | 2
Constipation (Gastrointestinal disorders) | 0 | 1 | 2
Diarrhea (Gastrointestinal disorders) | 0 | 2 | 6
Gastrointestinal disorders (Gastrointestinal disorders) | 0 | 0 | 1
Hemorrhoiids (Gastrointestinal disorders) | 0 | 1 | 2
Nausea (Gastrointestinal disorders) | 3 | 2 | 5
Proctitis (Gastrointestinal disorders) | 1 | 0 | 0
Rectal hemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Rectal pain (Gastrointestinal disorders) | 1 | 0 | 0
Salivary duct inflammation (Gastrointestinal disorders) | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 3
Edema limbs (General disorders) | 1 | 0 | 1
Fatigue (General disorders) | 3 | 1 | 4
Pain (General disorders) | 2 | 2 | 4
Upper respiratory infection (Infections and infestations) | 1 | 0 | 0
ry tract infection (Infections and infestations) | 1 | 0 | 0
Lymphocyte count decreased (Investigations) | 1 | 0 | 0
Neutrophil count decreased (Investigations) | 1 | 0 | 1
Platelet count decreased (Investigations) | 0 | 0 | 2
Weight loss (Investigations) | 0 | 0 | 2
White blood cell decreased (Investigations) | 2 | 2 | 3
Anorexia (Metabolism and nutrition disorders) | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 1
Hypokalemia (Metabolism and nutrition disorders) | 0 | 1 | 2
Hyponatremia (Metabolism and nutrition disorders) | 0 | 1 | 2
Avascular necrosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 1 | 0
Cystitis noninfective (Renal and urinary disorders) | 1 | 0 | 2
Renal and urinary disorders (Renal and urinary disorders) | 1 | 0 | 1
Urinary frequency (Renal and urinary disorders) | 1 | 1 | 1
Urinary incontinence (Renal and urinary disorders) | 0 | 1 | 1
Urinary tract pain (Renal and urinary disorders) | 1 | 0 | 0
Urinary urgency (Renal and urinary disorders) | 2 | 1 | 1
Dyspareunia (Reproductive system and breast disorders) | 0 | 1 | 4
Pelvic pain (Reproductive system and breast disorders) | 1 | 1 | 1
Vaginal hemorrhage (Reproductive system and breast disorders) | 1 | 0 | 0
Vaginismus (Reproductive system and breast disorders) | 1 | 0 | 0
Skin and subcutaneous tissue disorders (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Hot flashes (Vascular disorders) | 0 | 1 | 0
Lymphedema (Vascular disorders) | 0 | 0 | 1
Thromboembolic event (Vascular disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-12-03): https://cdn.clinicaltrials.gov/large-docs/88/NCT01627288/Prot_SAP_000.pdf